CLINICAL TRIAL: NCT02399774
Title: Dental Support Device During Breastfeeding as a Mean for Pain Control
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yariv yogev (Other)
Responsible Party: Sponsor-Investigator, Yariv yogev, Yariv Yogev, professor Director, division of obstetrics and delivery ward, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0087-15-RMC
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-03

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post-partum primi and multiparous women (Experimental): Post-partum primipara and multiparous women whom are interested in breastfeeding and have not begun yet. This arm will be randomized into 2 groups
  1. Intervention group: participants will receive the dental device and be instructed to use it during breastfeeding.
  2. Control group: participants will not receive any device for breastfeeding pain control
  Interventions: Device: Leboride
- Post-partum women that have already begun breast feeding (Experimental): 2. Post-partum women that have already begun breast feeding, will receive the dental device and each woman will be serve as her own control (breastfeeding before and after the use of the dental device.
  Interventions: Device: Leboride

INTERVENTIONS:
Device: Leboride — 1. Post-partum primi and multiparous women whom are interested in breastfeeding and have not begun yet. This arm will be randomized into 2 groups
     1. Intervention group: participants will receive the dental device and be instructed to use it during breastfeeding.
     2. Control group: participants will not receive any device for breastfeeding pain control
  2. Post-partum women that have already begun breast feeding, will receive the dental device and each woman will be serve as her own control (breastfeeding before and after the use of the dental device.

SUMMARY:
Leboride is a dental support device that was developed for reducing pain during active labor. It is made of an inert material, placed in the woman's mouth and does not disturb breathing, talking, or any other activity expected during labor. It is a single-use device, each user receives a new one.

This study hypothesis is that the Leboride use can reduce pain during breastfeeding, by that improve women's breastfeeding experience, and increase breastfeeding rates.

DETAILED DESCRIPTION:
Dental support device is effective in increasing isometric force in different muscle contraction [1-7]. In 2009 an avant-garde study [8] found in a small cohort that dental support device during labor, can shorten the second stage and reduce obstetrical interventions such as operative delivery and cesarean section. In this stage the woman has to contract muscles in order to push the fetus through the birth canal.

Leboride is a dental support device that was developed for reducing pain during active labor. It is made of an inert material, placed in the woman's mouth and does not disturb breathing, talking, or any other activity expected during labor. It is a single-use device, each user receives a new one.

This study hypothesis is that the Leboride use can reduce pain during breastfeeding, by that improve women's breastfeeding experience, and increase breastfeeding rates.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age 18-45 years.
2. Normal vital signs.

Exclusion Criteria:

1. Contraindications for breastfeeding.
2. Significant systemic disease that cause pain or require chronic pain relief.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1500 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Rate of change in of the vas scores before and after using this device | 24 months

SECONDARY OUTCOMES:
Duration of breastfeeding | 24 months
The rate of cessation of breastfeeding because of pain | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Director, Division of obstetrics and delivery
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel, Israel

REFERENCES:
- [Derived] Deussen AR, Ashwood P, Martis R, Stewart F, Grzeskowiak LE. Relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD004908. doi: 10.1002/14651858.CD004908.pub3. PMID 33078388